CLINICAL TRIAL: NCT05998187
Title: Mechanisms of Action on Rectal Motricity of Intrarectal Botulinum Toxin Injections in Patients With Fecal Incontinence
Brief Title: Mechanisms of Action on Rectal Motricity of Intrarectal Botulinum Toxin Injections
Acronym: MECA-TOX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/0384/HP
Record Dates: First submitted 2023-08-02; First posted 2023-08-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: Single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intra-rectal botulinum toxin injections (Experimental): Patients with fecal incontinence who have failed conservative treatments and are candidates for intra-rectal botulinum toxin injections.
  Interventions: Drug: intra-rectal botulinum toxin injections

INTERVENTIONS:
Drug: intra-rectal botulinum toxin injections — Patients with fecal incontinence who have failed conservative treatments and are candidates for intra-rectal botulinum toxin injections.

SUMMARY:
Previous studies have demonstrated the efficacy of this treatment in certain patients suffering from fecal incontinence, but it is not yet reimbursed in this indication as it is still in the evaluation phase. Indeed, little is known about botulinum toxin mechanisms of action. The aim of this study is to better understand the mechanisms of action of intra-rectal botulinum toxin injections, so that the investigators can identify the patients most likely to benefit from this treatment in the future.

DETAILED DESCRIPTION:
Fecal incontinence is a common condition, affecting around 5 to 6% of general population. Although not a serious condition, it severely impairs quality of life and leads to social isolation. Fecal incontinence also has a significant medico-economic cost. When first-line medical treatments fail (transit-regulating therapies, perineal re-education), fecal incontinence patients can be offered treatment with sacral nerve neuromodulation. However, this therapy will only be effective in the long term, and in terms of intention to treat, in less than half of patients who have had the device definitively implanted. Today, no other treatments are available apart from sphincter repair, for which the indications are very limited, or colostomy.

The investigator's team has therefore developed another therapeutic option, intra-rectal injections of botulinum toxin, in patients suffering from active fecal incontinence (i.e., preceded by defecatory urgency). The investigator have conducted two pilot studies, which demonstrated the efficacy of this treatment in an open-label setting, and the investigator are currently completing a randomized, double-blind, controlled study to confirm its efficacy (PHRCN 2014-003650-14). Nevertheless, the mechanisms of action of intra-rectal botulinum toxin injections remain hypothetical. By analogy with the intra-detrusor injections used for over 20 years to treat overactive bladder disease, it is possible that the toxin plays an inhibitory role on rectal motricity. Botulinum toxin inhibits the release of acetylcholine at the neuromuscular junction. Without this release, smooth muscle contraction cannot take place. In one of the two pilot, intra-rectal injections of botulinum toxin were performed in 6 patients with fecal incontinence and hyperactivity of the rectum or colonic reservoir after resection. In addition to the clinically demonstrated effect of these injections, there was a significant reduction in the amplitude of rectal contractions after injection. However, there was no correlation between the observed motor effect of botulinum toxin and the efficacy of the injections. Moreover, some patients did not exhibit colonic or rectal hypermotricity and still benefited from the injections. The investigator would like to continue exploring the motor effect of intra-rectal toxin injections on a larger group of patients suffering from faecal incontinence, using a more powerful motor recording system than anorectal manometry.

For this work, we hypothesize that intra-rectal botulinum toxin injections act primarily via a motor effect by inhibiting propagated rectal contractions. To test this hypothesis, a high-resolution recto-sigmoid manometry probe will be used to evaluate rectal and sigmoidal motricity spontaneously and in response to stimulant laxative injection, before and after intra-rectal injection of botulinum toxin. Patients included will be those suffering from faecal incontinence who have failed conservative treatments and are candidates for intra-rectal injections of botulinum toxin.

ELIGIBILITY:
Inclusion Criteria:

* Active or predominantly active fecal incontinence with failure of 1st-line conservative treatments (normalization of transit, perineal re-education)
* Impairment of quality of life at investigator's discretion
* Patients at least 18 years of age
* Patients who have read and understood the information letter and signed the consent form
* Patients affiliated to the French Social Security system
* Women of childbearing age using effective contraception (Cf. CTFG) (estro- progestins or intrauterine device or tubal ligation) for at least 1 month and a negative B-HCG urine pregnancy test at inclusion and for the duration of the study.
* Postmenopausal women: confirmatory diagnosis (non-medically induced amenorrhea for at least 12 months prior to inclusion visit)

Exclusion Criteria:

General

* Pregnant women, women in labor, breastfeeding women, or women without proven contraception
* Patient deprived of liberty by administrative or judicial decision, or protected adult (under guardianship or trusteeship)
* Exclusive passive fecal incontinence
* Patient suffering from constipation (Rome IV criteria)
* Patient with an evolving inflammatory or cancerous digestive pathology
* Previous rectal surgery
* Person participating in another research protocol or having participated in another research protocol in the 4 weeks preceding the inclusion visit

Linked to botulinum toxin injections

* Hypersensitivity to botulinum toxin or to one of the excipients (human albumin, sodium chloride)
* Neuromuscular junction pathology (myasthenia, Lambert-Eaton syndrome, etc.)
* Presence of infection at injection site(s)
* General anesthesia less than one month ago
* Association with aminoglycosides and anti-cholinesterase agents (risk of increased toxin effects)
* History of neurogenic damage such as polyradiculoneuritis
* History of dysphagia with esophageal or neurological stasis, swallowing disorders, inhalation pneumonitis
* Botulinum toxin injections in the 3 months preceding the study
* Clinical anal examination suggestive of anorectal abscess
* Recent history (<12 months) of myocardial infarction and/or rhythm disorders not reduced by appropriate treatment
* Peripheral motor neuropathies (such as amyotrophic lateral sclerosis or motor neuropathy) and underlying neurological disorders
* Current treatment with anticoagulants or anti-aggregants or haemostasis disorders according to recommendations (SFED). When patients are on anticoagulant or anti-aggregant therapy, the type of injections to be performed depends on the type of anticoagulation and the patient's thrombo-embolic risk:
* Patients on anticoagulant or anti-aggregant therapy with a major thrombo-embolic risk will not be included.
* Patients on anticoagulant or anti-aggregant therapy with a moderate or low thrombo-embolic risk may be included. If patients are taking a vitamin K antagonist, treatment will be continued provided that the INR is within the usual range of 2 to 3 (GETED, HAS, 2008). If patients are taking anti-aggregants, these can be continued (SFED, HAS, 2012). If patients are taking new oral anticoagulants, they should take a short break and not take the AOD the evening before or the morning of the injections (GIHP, 2015).

Linked to rectosigmoidoscopy

* Local pathology preventing colonoscopy (anal stenosis)
* Allergy or hypersensitivity to silicone and/or latex

Linked to laxatives

* Contraindication to DULCOLAX® 5 mg, gastro-resistant coated tablet
* Contraindication to XIMEPEG®, powder for oral solution

Linked to high-resolution manometry

* Clinically diagnosed intestinal obstruction
* Severe coagulopathy or oral anticoagulants
* Cardiac disorders for which vagal stimulation is poorly tolerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
high amplitude propagative contractions | before and 1 month after intrarectal botulinum toxin injections.
  The primary endpoint is the time to onset of high amplitude propagative contractions (HAPC) after instillation of DULCOLAX® in the sigmoid and rectum, before and 1 month after intrarectal botulinum toxin injections.

SECONDARY OUTCOMES:
Characteristics of contractions in the rectum and sigmoid | before and 1 month after intrarectal botulinum toxin injections.
  Amplitude of contractions in the rectum and sigmoid
Probe expulsion | before and 1 month after intrarectal botulinum toxin injections.
  Probe expulsion (which is an indirect sign of colorectal motricity efficiency) and time to probe expulsion.
Anal incontinence severity score | before and 1 month after botulinum toxin injections.
  Anal incontinence severity score (Cleveland Score) and stool schedule before and 1 month after botulinum toxin injections.
Quality of life score | before and 1 month after botulinum toxin injections.
  Quality of life score (FIQL Score, Appendix 4) before and 1 month after botulinum toxin injections.
Adverse events | at each visit, during 4 months
  Adverse events will be collected at each visits

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte DESPREZ, Principal Investigator — University Hospital, Rouen
Locations (1):
- Univesity Hospital, Rouen, Rouen, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao SS, Bharucha AE, Chiarioni G, Felt-Bersma R, Knowles C, Malcolm A, Wald A. Functional Anorectal Disorders. Gastroenterology. 2016 Mar 25:S0016-5085(16)00175-X 10.1053/j.gastro.2016.02.009. doi: 10.1053/j.gastro.2016.02.009. Online ahead of print. PMID 27144630
- [Background] Xu X, Menees SB, Zochowski MK, Fenner DE. Economic cost of fecal incontinence. Dis Colon Rectum. 2012 May;55(5):586-98. doi: 10.1097/DCR.0b013e31823dfd6d. PMID 22513438
- [Background] Desprez C, Damon H, Meurette G, Mege D, Faucheron JL, Brochard C, Lambrescak E, Gourcerol G, Mion F, Wyart V, Sielezneff I, Siproudhis L, Etienney I, Ajamie N, Lehur PA, Duflot T, Bridoux V, Leroi AM; Club NEMO. Ten-year Evaluation of a Large Retrospective Cohort Treated by Sacral Nerve Modulation for Fecal Incontinence: Results of a French Multicenter Study. Ann Surg. 2022 Apr 1;275(4):735-742. doi: 10.1097/SLA.0000000000004251. PMID 32740249
- [Background] Bridoux V, Gourcerol G, Kianifard B, Touchais JY, Ducrotte P, Leroi AM, Michot F, Tuech JJ. Botulinum A toxin as a treatment for overactive rectum with associated faecal incontinence. Colorectal Dis. 2012 Mar;14(3):342-8. doi: 10.1111/j.1463-1318.2011.02585.x. PMID 21689287
- [Background] Gourcerol G, Benard C, Melchior C, Touchais JY, Ducrotte P, Menard JF, Bridoux V, Leroi AM. Botulinum toxin: an endoscopic approach for treating fecal incontinence. Endoscopy. 2016 May;48(5):484-8. doi: 10.1055/s-0034-1393242. Epub 2015 Oct 8. PMID 26448532